CLINICAL TRIAL: NCT06529029
Title: Efficacy of Low Amplitude Pulse Seizure Therapy Versus Standard Ultra-Brief Right Unilateral Electroconvulsive Therapy in Remission of Suicidal Ideation
Brief Title: Low Amplitude Pulse Seizure Therapy Versus Standard Ultra-Brief Right Unilateral Electroconvulsive Therapy
Acronym: LAP-ST vs ECT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Pine Rest Christian Mental Health Services (Other)
Responsible Party: Principal Investigator, Nagy Youssef, MD, PhD, Vice President for Research; Director of Psychiatry and Behavioral Medicine Division -West Michican, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00010089
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Suicidal Ideation; Major Depressive Disorder; Schizo Affective Disorder; Bipolar Disorder
Keywords: Suicidal Ideation; Suicide; Depression; Major Depressive Disorder; Schizo Affective Disorder; Bipolar Disorder; Low Amplitude Seizure Therapy; Electroconvulsive Therapy; Neuromodulation; Brain Stimulation
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major; Psychotic Disorders; Bipolar Disorder; Suicide; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RUL LAP-ST (Low-Amplitude Pulse Seizure Therapy - Right Unilateral) (Experimental): Low Amplitude Pulse Seizure Therapy RUL ECT at 600mA (or 700mA)
  Interventions: Device: Sigma-Stim
- RUL ECT (Electroconvulsive Therapy) (Active Comparator): RUL Conventional pulse amplitude Electroconvulsive Therapy (ECT)
  Interventions: Device: Sigma-Stim

INTERVENTIONS:
Device: Sigma-Stim — Right Ultra-Brief Low Amplitude Seizure Therapy at 600mA or 700mA vs Right Unilateral Ultra-Brief Standard ECT at 800mA.

SUMMARY:
This protocol proposes an initial randomized clinical trial that includes all patients with suicidal ideation (SI) at baseline, and with SI as the primary outcome measure to examine whether Right Unilateral Low-Amplitude Pulse - Seizure Therapy (RUL LAP-ST) treatment has more magnitude and rate of remission of SI as conventional pulse amplitude Right Unilateral Electroconvulsive Therapy (RUL ECT) (based on our prior secondary analysis). Our central hypothesis is that RUL LAP-ST has significantly less cognitive/memory side effects (no memory side effects were noted in our prior studies for 500mA and 600mA) and thus is more favorable in terms of side effects compared to RUL conventional pulse amplitude ECT, while maintaining better anti-suicidal effect.

DETAILED DESCRIPTION:
Suicide is one of the leading causes of mortality. Suicidal Ideation (SI) is a precursor to suicide. SI is especially hard to treat/remit in those with treatment-resistant psychiatric disorders (TRPD). This includes treatment-resistant mood disorders and psychotic disorders (such as schizophrenia and schizoaffective disorders). The above TRPD and the SI can remit with Electroconvulsive Therapy (ECT). That is to say, a transdiagnostic, evidence-based treatment for those patients, in addition to pharmacotherapy and psychotherapy, is ECT. ECT has both research support (mainly secondary analysis) and clinical evidence of a beneficial effect in remission of suicidality, as well as unsurpassed effect in treating primary mood and psychotic disorders including those who are treatment-resistant to other therapeutics. However, there are undeniable barriers to treatment with ECT. The most important barrier is memory side effects. ECT can help SI. ECT has also been shown to improve quality of life in a randomized trial by our group, which studied elderly patients with depression. Treating SI, along with the underlying disorder, especially in patients with TRPD is crucial in real-world patients who are clinically referred for ECT. These real-world referrals to ECT (by the patients' primary psychiatrist) will constitute the recruitment pool for this study.

Current amplitude drives electric fields to the deeper structures that are concerned with memory (Peterchev et al., 2010). Previously, the investigators performed the first in human proof of concept one arm open label clinical trial of LAP-ST, (N=22); followed by another small (N=7) pilot randomized, double-blinded clinical trial for the feasibility, safely and initial efficacy of LAP-ST, and another group later confirmed the more favorable cognitive side effects of LAP-ST compared to higher current amplitude (800mA).

However, efficacy of LAP-ST against suicidality has not been well established as primary outcome previously.

Thus, this protocol proposes an initial randomized clinical trial that includes all patients with SI at baseline, and with SI as the primary outcome measure to examine whether RUL LAP-ST treatment has more magnitude and rate of remission of SI as conventional pulse amplitude RUL ECT (based on our prior secondary analysis). Our central hypothesis is that RUL LAP-ST has significantly less cognitive/memory side effects (no memory side effects were noted in our prior studies for 500mA or 600mA) and thus is more favorable in terms of side effects compared to RUL conventional pulse amplitude ECT, while maintaining better anti-suicidal effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom ECT is clinically indicated: The referrals to ECT by the primary psychiatrist (before a consult by the ECT consultant) will serve to both increase the feasibility of the study and address any ethical concerns that the patient would not undergo ECT without having a valid full indication for the procedure as well as increase the external validity and generalizability of the study.
2. Male or female patients 18 to 90 years of age
3. Current DSM-5 criteria for MDE with any SI of major depressive, bipolar, or schizoaffective disorders
4. Montgomery-Asberg depression rating scale (MADRS) with 2 or more on SI item
5. Use of effective method of birth control for women of child-bearing capacity
6. Patient is medically stable
7. No anticipated need to alter psychotropic medications for the duration of the study (except for urgent/emergent situations)
8. Ability of patient to fully participate in the informed consent process

Exclusion Criteria:

1. Unstable or serious medical condition that substantially increases risks of ECT or cognitive impairment
2. Female patients who are pregnant or plan to be pregnant during the study or are breast-feeding
3. History of neurological disorder if deemed by the treating ECT physician or PI to pose a significant risk with ECT, or if there is any metal in the head or history of known structural brain lesion or skull defect that is deemed to affect cognition or safe ECT treatment
4. Implanted devices that make ECT unsafe
5. Clinical presentation of delirium or dementia
6. Active substance use disorders within 1 week of randomization
7. ECT in the past 1 month or prior failure to respond to an adequate course of ECT as deemed by the ECT physician treating the patient or the PI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Suicide Ideation - Self Report | Through study completion, an average of four weeks
  Beck Scale for Suicide Ideation (SSI-Worst and SSI-Current) - self reported. Minimum score of 0, maximum score of 42. Lower score indicates a better outcome.
Suicide Ideation - Clinician Rated | Through study completion, an average of four weeks
  Columbia Suicide Severity Rating Scale (C-SSRS) - clinician administered. Intensity of suicidal ideation: minimum score of 0, maximum score of 5. Lower score indicates a better outcome. Suicidal behavior not rated on a scale.

SECONDARY OUTCOMES:
Depression - Clinician Rated | Through study completion, an average of four weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) - clinician administered. Minimum score of 0, maximum score of 60. Lower score indicates better outcome.
Depression - Self Report | Through study completion, an average of four weeks
  Patient Health Questionnaire (PHQ9) - self reported. Minimum score of 0, maximum score of 27. Lower score indicates better outcome.
Depression - Self Report | Through study completion, an average of four weeks
  Quick Inventory of Depressive Symptomatology (QIDS-SR) - self reported. Minimum score of 0, maximum score of 27. Lower score indicates better outcome.

OTHER OUTCOMES:
Anxiety | Through study completion, an average of four weeks
  Generalized Anxiety Disorder (GAD7) - self reported. Minimum score 0, maximum score 21. Lower score indicates better outcome.
Psychosis | Through study completion, an average of four weeks
  Positive and Negative Syndrome Scale (PANSS) - clinician administered. Full scale minimum score of 31. Maximum score of 217. Lower score indicates better outcome.
Global Clinical Assessment | Through study completion, an average of four weeks
  Clinical Global Improvement (CGI) - clinician administered. Severity: minimum score of 0, maximum score of 7, lower score indicates better outcome. Improvement: minimum score of 0, maximum score of 7, lower score indicates better outcome.
Time to Reorientation after ECT sessions | Through study completion, an average of four weeks
  Time to Reorientation scale (TRO) - study staff administered. Minimum score 3 minutes, maximum score more than 20 minutes. Lower score indicates better outcome.
Cognitive function and cognitive side effects | At baseline and completion of the acute ECT/LAP-ST course, an average of four weeks
  Hopkins Verbal Learning Test-Revised (HVLTR) - clinician administered. Minimum score of 0, maximum score of 12. Higher score indicates better outcome.
Cognitive Executive functions | At baseline and completion of the acute ECT/LAP-ST course, an average of four weeks
  Delis Kaplan Executive Function Scale (DKEFS) - verbal fluency and color/word interference modules - clinician administered. Verbal fluency: minimum score of 1, maximum score of 60. Higher scores indicate better outcome for the total score. Color-word interference: minimum score of 1, maximum score of 19. In general, higher score indicate better outcome.
Autobiographic Memory side effects | At baseline and completion of the acute ECT/LAP-ST course, an average of four weeks
  Autobiographic Memory Interview-Short Form (AMI-SF) - clinician administered. Minimum score of 0, maximum score of 30. Higher score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nagy A Youssef, MD, PhD, Principal Investigator — Pine Rest Christian Mental Health Services & Michigan State University
Locations (1):
- Pine Rest Christian Mental Health Services, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kochanek KD, Murphy S, Xu J, Arias E. Mortality in the United States, 2016. NCHS Data Brief. 2017 Dec;(293):1-8. PMID 29319473
- [Background] Curtin S, Warner M, Hedegaard H: Increase in suicide in the United States, 1999-2014. NCHS data brief no. 241. Hyattsville, MD: US Department of Health and Human Services, CDC, National Center for Health Statistics. https://www.cdc.gov/nchs/data/databriefs/db241.pdf. 2016
- [Background] Kellner CH, Fink M, Knapp R, Petrides G, Husain M, Rummans T, Mueller M, Bernstein H, Rasmussen K, O'connor K, Smith G, Rush AJ, Biggs M, McClintock S, Bailine S, Malur C. Relief of expressed suicidal intent by ECT: a consortium for research in ECT study. Am J Psychiatry. 2005 May;162(5):977-82. doi: 10.1176/appi.ajp.162.5.977. PMID 15863801
- [Background] Fink M, Kellner CH, McCall WV. The role of ECT in suicide prevention. J ECT. 2014 Mar;30(1):5-9. doi: 10.1097/YCT.0b013e3182a6ad0d. PMID 24091903
- [Background] Sienaert P. Based on a True Story? The Portrayal of ECT in International Movies and Television Programs. Brain Stimul. 2016 Nov-Dec;9(6):882-891. doi: 10.1016/j.brs.2016.07.005. Epub 2016 Jul 20. PMID 27522170
- [Background] McCall WV, Lisanby SH, Rosenquist PB, Dooley M, Husain MM, Knapp RG, Petrides G, Rudorfer MV, Young RC, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Youssef NA, McCloud L, Kellner CH; CORE/PRIDE Work Group. Effects of continuation electroconvulsive therapy on quality of life in elderly depressed patients: A randomized clinical trial. J Psychiatr Res. 2018 Feb;97:65-69. doi: 10.1016/j.jpsychires.2017.11.001. Epub 2017 Nov 16. PMID 29195125
- [Background] Kulak-Bejda A, Bejda G, Waszkiewicz N. Mental Disorders, Cognitive Impairment and the Risk of Suicide in Older Adults. Front Psychiatry. 2021 Aug 25;12:695286. doi: 10.3389/fpsyt.2021.695286. eCollection 2021. PMID 34512415
- [Background] Lara E, Olaya B, Garin N, Ayuso-Mateos JL, Miret M, Moneta V, Haro JM. Is cognitive impairment associated with suicidality? A population-based study. Eur Neuropsychopharmacol. 2015 Feb;25(2):203-13. doi: 10.1016/j.euroneuro.2014.08.010. Epub 2014 Aug 21. PMID 25190638
- [Background] Fernandez-Sevillano J, Alberich S, Zorrilla I, Gonzalez-Ortega I, Lopez MP, Perez V, Vieta E, Gonzalez-Pinto A, Saiz P. Cognition in Recent Suicide Attempts: Altered Executive Function. Front Psychiatry. 2021 Jul 22;12:701140. doi: 10.3389/fpsyt.2021.701140. eCollection 2021. PMID 34366931
- [Background] Rutter SB, Cipriani N, Smith EC, Ramjas E, Vaccaro DH, Martin Lopez M, Calabrese WR, Torres D, Campos-Abraham P, Llaguno M, Soto E, Ghavami M, Perez-Rodriguez MM. Neurocognition and the Suicidal Process. Curr Top Behav Neurosci. 2020;46:117-153. doi: 10.1007/7854_2020_162. PMID 32860213
- [Background] Szanto K, Galfalvy H, Vanyukov PM, Keilp JG, Dombrovski AY. Pathways to Late-Life Suicidal Behavior: Cluster Analysis and Predictive Validation of Suicidal Behavior in a Sample of Older Adults With Major Depression. J Clin Psychiatry. 2018 Mar/Apr;79(2):17m11611. doi: 10.4088/JCP.17m11611. PMID 29489076
- [Background] Deng ZD, Lisanby SH, Peterchev AV. Electric field strength and focality in electroconvulsive therapy and magnetic seizure therapy: a finite element simulation study. J Neural Eng. 2011 Feb;8(1):016007. doi: 10.1088/1741-2560/8/1/016007. Epub 2011 Jan 19. PMID 21248385
- [Background] Peterchev AV, Rosa MA, Deng ZD, Prudic J, Lisanby SH. Electroconvulsive therapy stimulus parameters: rethinking dosage. J ECT. 2010 Sep;26(3):159-74. doi: 10.1097/YCT.0b013e3181e48165. PMID 20805726
- [Background] Youssef N, Sidhom E: Examination of Cognitive Profile and Variability in the Current Amplitude Domain of Low Current Amplitude ECT in Society of Biological Psychiatry 69th Annual Meeting (Published in Biological Psychiatry 2014 supplement) New York, New York2014
- [Background] Youssef NA, Sidhom E. Feasibility, safety, and preliminary efficacy of Low Amplitude Seizure Therapy (LAP-ST): A proof of concept clinical trial in man. J Affect Disord. 2017 Nov;222:1-6. doi: 10.1016/j.jad.2017.06.022. Epub 2017 Jun 16. PMID 28667887
- [Background] Youssef NA, McCall WV, Ravilla D, McCloud L, Rosenquist PB. Double-Blinded Randomized Pilot Clinical Trial Comparing Cognitive Side Effects of Standard Ultra-Brief Right Unilateral ECT to 0.5 A Low Amplitude Seizure Therapy (LAP-ST). Brain Sci. 2020 Dec 13;10(12):979. doi: 10.3390/brainsci10120979. PMID 33322138
- [Background] Youssef NA, Ravilla D, Patel C, Yassa M, Sadek R, Zhang LF, McCloud L, McCall WV, Rosenquist PB. Magnitude of Reduction and Speed of Remission of Suicidality for Low Amplitude Seizure Therapy (LAP-ST) Compared to Standard Right Unilateral Electroconvulsive Therapy: A Pilot Double-Blinded Randomized Clinical Trial. Brain Sci. 2019 Apr 29;9(5):99. doi: 10.3390/brainsci9050099. PMID 31035665
- [Background] Abbott CC, Quinn D, Miller J, Ye E, Iqbal S, Lloyd M, Jones TR, Upston J, Deng Z, Erhardt E, McClintock SM. Electroconvulsive Therapy Pulse Amplitude and Clinical Outcomes. Am J Geriatr Psychiatry. 2021 Feb;29(2):166-178. doi: 10.1016/j.jagp.2020.06.008. Epub 2020 Jun 17. PMID 32651051
- [Background] Beck AT, Brown GK, Steer RA. Psychometric characteristics of the Scale for Suicide Ideation with psychiatric outpatients. Behav Res Ther. 1997 Nov;35(11):1039-46. doi: 10.1016/s0005-7967(97)00073-9. PMID 9431735
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082